CLINICAL TRIAL: NCT03522857
Title: Measuring Healthcare Professional Students Knowledge and Attitudes Towards Chronic Pain Management.
Brief Title: Healthcare Professional Students' Knowledge and Attitudes Towards Chronic Pain Management.
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: King's College London (Other); Glasgow Caledonian University (Other); University of Nottingham (Other); Northumbria University (Other); Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Principal Investigator, Teesside University
Other Study IDs: SA 144/17
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Chronic Pain; Student Education; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Chronic Pain; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Teesside University: nursing, midwifery, physiotherapy, occupational therapy, diagnostic radiography, paramedics
- Glasgow Caledonian University: nursing, midwifery, physiotherapy, occupational therapy, diagnostic radiography, paramedics
- Northumbria University: nursing, midwifery, physiotherapy, occupational therapy
- University of Nottingham: Physiotherapy, nursing and midwifery
- Curtin University: Physiotherapy
- Notre Dame University: Physiotherapy
- University College Dublin: Physiotherapists
- Leeds Beckett University: Physiotherapists
- University College Cork: Physiotherapists
- Robert Gordon University: OT, Physio, Midwifery, Nursing, Diagnostic radiography
- University of Ulster: Physiotherapy
- University of Limerick: OT, Physio, Midwifery, Nursing, Diagnostic radiography, paramedic

SUMMARY:
Chronic pain affects from one third to one half of the population in the UK (Fayaz et al, 2016). The cost and burden of chronic pain is significant to health services worldwide. The affects of chronic pain are widespread upon the lives of those affected. Health professionals need to be better equipped than at present to manage pain and current chronic pain management knowledge in healthcare is poor. Briggs et al 2011 described the hours of pain education delivered at undergraduate level as 'woefully inadequate'. The International Association for Study of Pain (IASP) defined curricula for pain education at undergraduate level 6 years ago but current levels of knowledge at undergraduate health professional level are not widely known. This study aims to establish this at the outset of a pre-registration health professional courses and at the end of these courses.

This study aims to identify the baseline knowledge and attitudes of pre-registration healthcare students in Universities throughout UK and Ireland toward chronic pain management. The disciplines targeted are nursing, midwifery, physiotherapy, occupational therapy, diagnostic radiography and paramedics.

It is a cross sectional study that compares attitudes and knowledge of first year and final year pre-registration healthcare students in the UK and Ireland. These parameters are measured using the HC-PAIRS measure and Revised Neurophysiology Questionnaire respectively. In addition anonymous data is collected pertaining to participant characteristics which are institute of study, age, gender, level and discipline of study to enable a comparison between these parameters.

DETAILED DESCRIPTION:
Chronic pain is characterised by a protective mechanism of the neuro-immune-endocrine systems potentially exacerbated by loading exposures, conditioning, psychological, socio-economic, lifestyle, comorbid mental health and non-modifiables such as genetics, (O'Sullivan et al 2016). Pain education can be a useful basis for helping patients to manage their symptoms and return to good daily function. However a biomedical approach to chronic pain persists in medical communities, whilst persistent pain populations increase and incidences of opioid addiction are growing secondary to poor pain management. Biomedical models of pain are likely to induce fear avoidant behaviour and exacerbate chronicity (Wertli et al 2014). In order to change the prevailing biomedical approach to chronic pain the International Association for the Study of Pain (IASP) have provided detailed pain curricula content for different medical and allied health professional courses. Briggs et al (2015) found that out of 15 'representative European countries' less than a handful of universities from 3 countries had implemented distinctly identifiable pain education teaching. However they may be other forms of pain education that are taking place in pre-registration healthcare professional education. This study aims to establish the levels of chronic pain management knowledge and attitudes prevail in the UK and Ireland amongst pre-registration healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

- pre-registration healthcare student, BSc or MSc.

Exclusion Criteria:

- post-registration students

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: University students in UK and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Revised Neurophysiology Quiz | 1 day
  12 point pain knowledge quiz devised originally by Moseley 2003 to assess knowledge of biological mechanisms of pain. Revised and reduced in 2013 by Catley et al. The lowest score is 0 and the highest would be 12 on a scale of 0-12. There are no subscales.
Health care providers Pain and Impairment Relationship Scale | 1 day
  A 13 question, 7 point Likert scale and a validated questionnaire to assess health care providers' attitudes and beliefs about the relationship between pain and impairment. The scale ranges in outcome from 0-90, higher scores representing a stronger belief in the relationship between chronic pain and disability (a 'worse outcome') and lower scores representing a reduced belief on this relationship thus a 'better outcome'. There are no subscales.

SECONDARY OUTCOMES:
Biographic data | 1 day
  age in years
Biographic data (gender) | 1 day
  gender (male/female)
Biographic data (discipline) | 1 day
  discipline (nursing, midwifery, physiotherapy, occupational therapy, paramedics, diagnostic radiotherapy)
Biographic data (Degree qualification) | 1 day
  level of study (BSc/MSc)
Biographic data (stage of study) | 1 day
  Year of study (first or final year)
Biographic data (Institute) | 1 day
  University of study

CONTACTS AND LOCATIONS:
Overall Officials: Jagjit Mankelow, MSc, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

REFERENCES:
- [Derived] Mankelow J, Ryan CG, Taylor PC, Casey MB, Naisby J, Thompson K, McVeigh JG, Seenan C, Cooper K, Hendrick P, Brown D, Gibson W, Travers M, Kennedy N, O'Riordan C, Martin D. International, multi-disciplinary, cross-section study of pain knowledge and attitudes in nursing, midwifery and allied health professions students. BMC Med Educ. 2022 Jul 15;22(1):547. doi: 10.1186/s12909-022-03488-3. PMID 35840942